CLINICAL TRIAL: NCT07242495
Title: Additional Effects of Immersive vr 360 Degree Videos With Aerobic Exercises on Cognitive Functions in Elderly With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/09
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Dysfunctions; Cognitive Disorder; Cognitive Decline
Keywords: Cognitive rehabilitation; Virtual Reality; Mild cognitive Impairment; Elderly; Aerobic exercise
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR 360 degree Videos and Aerobic Chair Exercises intervention (Experimental): Intervention: Combination of immersive VR 360° videos and structured chair-based aerobic exercises Session Duration: Starts at 15 minutes, progresses up to 25 minutes Frequency: 2 sessions per week Total Duration: 6 weeks VR Content: Forest, wildlife, space, wildlife, solar system, waterfalls, room environments
  Aerobic Exercises: Chair-based aerobic exercises (upper and lower limb movements, rhythmic seated marching, arm raises) Additional Task: Short memory recall activity to explain the main events, details and characters in the VR 360 degree video at the end of each VR session
  Interventions: Procedure: VR 360 degree Videos and Aerobic Chair Exercises intervention
- Chair Aerobic Exercises (Active Comparator): Chair aerobic exercises 15 min/day with progression upto 25 min, 2 days a week, for 6 weeks.
  Chair aerobic exercise includes:
  1. Alternate heel digs with bilateral biceps curl 8 repetitions per session.
  2. V- Step with bilateral hammer curls 8 repetitions per session.
  3. Lateral step touch with bilateral biceps curls 8 repetitions per session.
  4. Knee lift 8 repetitions per session.
  5. Arm swings 8 repetitions per session.
  6. Clap swing 8 repetitions per session.
  7. Sit, stand and clap 8 repetitions per session
  Interventions: Procedure: Chair Aerobic Exercises

INTERVENTIONS:
Procedure: VR 360 degree Videos and Aerobic Chair Exercises intervention — Combination of immersive VR 360° videos and structured chair-based aerobic exercises Session Duration: Starts at 15 minutes, progresses up to 25 minutes Frequency: 2 sessions per week Total Duration: 6 weeks VR Content: Forest, wildlife, space, wildlife, solar system, waterfalls, room environments
  Aerobic Exercises: Chair-based aerobic exercises (upper and lower limb movements, arm raises) Additional Task: Short memory recall activity to explain the main events, details and characters in the VR 360 degree video at the end of each VR session.
  Arms: VR 360 degree Videos and Aerobic Chair Exercises intervention
Procedure: Chair Aerobic Exercises — Chair aerobic exercises 15 min/day with progression upto 25 min, 2 days a week, for 6 weeks.
  Chair aerobic exercise includes:
  1. Alternate heel digs with bilateral biceps curl 8 repetitions per session.
  2. V- Step with bilateral hammer curls 8 repetitions per session.
  3. Lateral step touch with bilateral biceps curls 8 repetitions per session.
  4. Knee lift 8 repetitions per session.
  5. Arm swings 8 repetitions per session.
  6. Clap swing 8 repetitions per session.
  7. Sit, stand and clap 8 repetitions per session
  Arms: Chair Aerobic Exercises

SUMMARY:
One of the key challenges faced by individuals with Mild Cognitive Impairment (MCI) is the decline in cognitive abilities, particularly global cognition, attention, and executive function, which are essential for maintaining independence and performing daily activities. Impaired cognition can significantly reduce quality of life in older adults, leading to difficulties in managing routine tasks, reduced social engagement, and increased dependency on caregivers. Common signs and symptoms include forgetfulness, difficulty concentrating, slower problem-solving, and challenges in planning or organizing daily activities. This study aims to explore and compare the effectiveness of two interventions-immersive Virtual Reality (VR) 360-degree videos combined with aerobic exercises, and aerobic exercises alone-in improving cognitive functions in older adults with MCI. Key outcome measures, including the Montreal Cognitive Assessment (MoCA) and Trail Making Test (TMT), will evaluate the effectiveness of the interventions on global cognition, attention, and executive function. We will include older adults aged 60 years and above with MoCA scores between 18-25 (MCI patients), who are able to perform independent ADLs. The participants will be assessed at the start of the intervention through the MoCA scale for MCI screening and baseline TMT testing for inclusion.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is a transitional stage between normal aging and dementia, characterized by a noticeable decline in cognitive abilities that does not yet significantly interfere with daily functioning. The prevalence of MCI in older adults is estimated to be around 15-20%, and individuals with this condition often face challenges in memory, attention, and executive function. These impairments can reduce independence, limit participation in daily activities, and increase the risk of progression to dementia or Alzheimer's disease. One of the major consequences of cognitive decline is difficulty in maintaining attention and executive control, which are essential for managing everyday tasks such as planning, organizing, and problem-solving. This decline not only affects quality of life but also places a greater burden on caregivers and healthcare systems.

Non-pharmacological interventions have gained increasing attention as pharmacological treatments have shown limited effectiveness in slowing the progression of MCI. Aerobic exercise has long been recognized for its positive effects on both physical and cognitive health, improving blood flow, neuroplasticity, and memory functions. More recently, immersive Virtual Reality (VR) 360-degree videos have emerged as a promising tool for cognitive rehabilitation. VR provides enriched sensory stimulation and engaging environments that can enhance attention, memory, and executive processes by immersing individuals in interactive and stimulating experiences.

This study aims to determine the additional effects of combining immersive VR 360-degree videos with aerobic exercises on cognitive functions in elderly individuals with MCI. By comparing two interventions-VR 360-degree videos with aerobic exercises versus aerobic exercises alone-this research seeks to evaluate whether VR can amplify the cognitive benefits of exercise. The intervention group will undergo a 6-week program consisting of VR 360-degree videos combined with aerobic exercises, starting with 15-minute sessions twice a week and progressing up to 25 minutes. The control group will perform chair-based aerobic exercises of the same duration and frequency without VR.

Key outcome measures, including the Montreal Cognitive Assessment (MoCA) and the Trail Making Test (TMT), will be used to assess global cognition, attention, and executive function. Assessments will be conducted at baseline, mid-point (3rd week), and post-intervention (6th week). Participants will be older adults aged 60 years and above with MoCA scores between 18-25, who are able to perform independent activities of daily living. Eligible participants will be recruited through non-probability convenient sampling and randomly assigned into two groups using the coin toss method.

This single-blinded randomized controlled trial will be conducted at Fauji Foundation Hospital, Rawalpindi, over the course of one year following ethical approval. By exploring the combined effects of VR and aerobic exercise, this study aims to provide valuable insights into innovative, accessible, and engaging interventions that can support cognitive health in older adults with MCI, ultimately improving their quality of life and delaying further cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Older population aged from 60years and above
* Normal/ normal to corrected vision
* MoCA Score of 18-25 for screening / MCI patients
* Can do Independent ADLS

Exclusion Criteria:

* Individuals with preexisting conditions such as severe motion sickness that could be exacerbated by VR usage.
* Communication impairments
* Participants with other neurological disorders.
* Sensory deficits (such as uncontrolled hearing or visual issues)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 6 weeks
  Montreal Cognitive Assessment (MoCA) will be used for this. Values:
  26-30 = Normal cognition 18-25 = Mild Cognitive Impairment (MCI) 10-17 = Moderate cognitive impairment
  <10 = Severe cognitive impairment
Attention | 6 weeks
  Trail Making Test will be used for this. Values:
  TMT-A:
  <40 seconds = Above average 40-60 seconds = Average
  TMT-B:
  <75 seconds = Above average 75-180 seconds = Average

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan